CLINICAL TRIAL: NCT03520049
Title: Proof of Concept; A Pilot, Randomized, Double-Blind Study of Oseltamivir Versus Placebo for Immune Thrombocytopenia
Brief Title: Proof-of-Concept: A Pilot, Randomized, Double-Blind Study of Oseltamivir Versus Placebo for Immune Thrombocytopenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Li Ka Shing Knowledge Institute (Unknown); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITP30
Record Dates: First submitted 2017-10-03; First posted 2018-05-09 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Immune Thrombocytopenia
Keywords: Thrombocytopenia; ITP; Platelets; Bleeding; Immune; Oseltamivir; Glycoprotein; Sialylation; Antibody; Autoantibody
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Hemorrhage | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oseltamivir (Experimental): Oseltamivir capsule administered orally at 75 mg twice daily for five consecutive days.
  Interventions: Drug: Oseltamivir
- Placebo (Placebo Comparator): Placebo capsule administered orally twice daily for five consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oseltamivir
  Other Names: Oseltamivir phosphate; Tamiflu®
  Arms: Oseltamivir
Drug: Placebo
  Arms: Placebo

SUMMARY:
Immune Thrombocytopenia (ITP) is a disorder resulting in impaired platelet production and enhanced destruction on the basis of autoantibody-mediated mechanisms. Patients with ITP are at increased risk of bleeding and infection. First line therapy includes glucocorticoids, with or without the addition of intravenous immune globulin (IVIg) when a prompt platelet response is desired. The likelihood of stable and safe disease after first-line treatment ranges from 30-60% and risk of relapse requiring additional therapy occurs in 50-80% of patients. Moreover, the toxicity associated with first and subsequent therapy for ITP is substantial.

Oseltamivir is an attractive drug for ITP since it specifically targets a pathophysiologic mechanism that appears to be important for the development of ITP and has a benign side effect profile compared to standard ITP therapy.

Oseltamivir has never been rigorously tested in humans to determine its efficacy in the management of ITP. The investigators therefore propose the first randomized, double blind study to assess the impact of oseltamivir on biological markers in adult patients with ITP. This study will also provide information about the feasibility of recruitment into a definitive trial, which would be coordinated by St. Michael's Hospital.

The research question is: Do adults (≥ 18 years) with ITP treated with oseltamivir at 75mg twice daily for 5 consecutive days have an increase in their mean platelet glycoprotein sialylation compared to those receiving placebo?

This pilot, proof-of-concept, randomized controlled clinical trial will enroll 30 individuals with ITP. Randomization and allocation will occur at a ratio of 1:1. Analysis of the primary outcome measure will occur via analysis of covariance (ANCOVA).

This study has the potential to dramatically change the treatment of ITP. If the results from this study demonstrate a biological effect, and results from the subsequent definitive study are positive, The investigators envision a move away from non-specific immune-blunting therapy such as prednisone, towards tailored therapy with oseltamivir. It could diminish the lifelong summative immunosuppressive therapy burden, associated drug toxicity and improve long- and short-term health outcomes for these patients.

DETAILED DESCRIPTION:
Explanation (of rationale for current study):

Despite the encouraging case report described above, oseltamivir has not been rigorously tested in humans to determine its efficacy in the management of ITP. Oseltamivir is an attractive drug for ITP since it specifically targets a pathophysiologic mechanism that appears to be important for the development of ITP and has a benign side effect profile compared to standard ITP therapy. However, more robust evidence that oseltamivir affects desialylation in humans is needed before a definitive, multicenter randomized trial can be justified to funders.

The investigators therefore propose the first randomized, double blind, study to assess the impact of oseltamivir on biological markers in adult patients with ITP. This study will also provide information about the feasibility of recruitment into a definitive trial, which would be coordinated at St. Michael's Hospital (SMH).

Impact:

The most appropriate treatment of patients with persistent ITP represents an area of major clinical interest burdened by unacceptable uncertainty. This study has the potential to dramatically change the treatment of ITP. If the results from the definitive study are positive, the investigators envision a move away from non-specific immune-blunting therapy such as prednisone, towards tailored therapy like oseltamivir. Targeted therapy for ITP is a timely and relevant concept. It could diminish the lifelong summative immunosuppressive therapy burden, associated drug toxicity and improve long- and short-term health outcomes for this patient population.

Research Question:

Do adults (≥ 18 years) with ITP treated with oseltamivir at 75mg twice daily for 5 consecutive days have an increase in their mean platelet glycoprotein sialylation compared to those receiving placebo?

Primary Objective:

The primary objective of this study is to assess the impact of oseltamivir on mean platelet glycoprotein sialylation when administered orally at 75 mg twice daily versus placebo for five consecutive days in the management of ITP in adult patients (≥ 18 years).

Secondary Objectives:

The secondary objectives relate to the feasibility of conducting a subsequent definitive randomized trial focused on treatment efficacy and include:

1. The percentage of eligible patients who were successfully recruited;
2. The number of patients recruited per month;
3. The percentage of patients who received the study drug within 12 hours of randomization;
4. The percentage of patients who received every scheduled dose of the study drug in a blinded fashion;
5. The percentage of patients who completed follow-up six months after randomization.

Additional exploratory objectives are to determine in each treatment arm:

1. The mean platelet count;
2. The proportion of patients who received additional ITP based therapy during the study 12 month follow-up period;
3. Frequencies of CD4+ and CD8+ T regulatory cells;
4. Cytokine profiles;
5. The anti-platelet glycoprotein antibody specificity/titer; and
6. The effects of these antibodies on macrophage- and hepatocyte-mediated Fc-dependent and independent phagocytosis in vitro.

Methods: Trial Design, Participants, Interventions, and Outcomes:

Trial Design:

This is a single center, pilot, proof-of-concept, double-blind randomized controlled clinical trial to determine the impact of oseltamivir on mean platelet glycoprotein sialylation in patients with ITP. Eligible participants will be randomized to one of two treatment regimens in a 1:1 allocation ratio, receiving either oseltamivir (administered orally at 75 mg twice daily) or placebo (administered orally twice daily) for five consecutive days.

Information for Participants:

Those who are capable of giving informed consent meeting study eligibility criteria, as per the investigators judgement, will be approached for study. The informed consent form (ICF) and process for obtaining informed consent will comply with institutional, local, national and international laws, rules and regulations. The ICF will be signed and dated by the subject before the subject participates in any study-related activities. If any significant changes to study design are made, a protocol amendment will be issued, submitted/approved by the REB and signed by the site investigator. Protocol changes will be presented to the subject and repeated ICF procedures will occur.

Study Site:

This will be a single center study undertaken at SMH, Toronto, Ontario, Canada. All laboratory based elements will be measured/studied at the SMH clinical hematology lab or at Dr. Ni's platelet biology lab at the Li Ka Shing Knowledge Institute.

Description of Interventions:

All study participants will receive either oseltamivir (administered orally at 75 mg twice daily) or placebo (administered orally twice daily) for five consecutive days. Screening of potential study participants will occur within 7 days of the randomization date (Day 0). Screening can occur on Day 0. The study participant will be randomized on Day 0 and study drug administration will begin on Day 1 and end on Day 5.

All capsules will be dispensed in a blister pack format. The capsules of oseltamivir and placebo will be encapsulated to look the same. Packing and labeling of the blister packs will be performed by the study pharmacist at SMH. To track compliance, the blister pack will be reviewed at Day 5 (or within 3 days of study drug completion) and a participant diary will be utilized. Discontinuation of the medication while on trial can occur because of adverse effects, participant or treating physician request (e.g. if patient requires standard ITP therapy). The reason for discontinuation will be carefully collected and documented. For the duration of the trial, there will be no additional study interventions aside from what has already been described above.

Co-Interventions:

The investigators anticipate that rare patients will receive additional ITP therapy over the course of study follow-up, particularly if their platelet count falls to below 20 x 109/L. Therefore, the investigators will collect data regarding immunosuppressive therapy at all follow-up time points.

Feasibility of Intervention and Study Population Oseltamivir is a safe and well-tolerated medication. The dose and duration of treatment used in this study is the accepted regimen for the treatment of influenza. The most common side effects (2-15%) are gastrointestinal symptoms (nausea, abdominal pain and diarrhea). Current second/third line management of ITP involves a range of immunosuppressive regimens with variable efficacy and considerable adverse effects, or observation without therapy (depending on a patient's platelet count and bleeding risk). The placebo and oseltamivir treatment arms are ethically sound for the reasons listed above and because the investigators are excluding patients with severe thrombocytopenia (<20 x E9/L) and active significant bleeding (defined as a bleeding assessment score of Grade 2 at any site by the Immune Thrombocytopenia Purpura Bleeding Score).

Methods: Randomization

Sequence Generation, Concealment of Allocation and Implementation:

Concealment of allocation will occur by centralized web based randomization using sealed envelopes, with a 1:1 computer generated allocation sequence created independently by the study statistician, Prof. Kevin Thorpe. Participants will be randomized with permuted blocks of varying size to achieve allocation balance across the two treatment groups (this will be concealed to participants, clinicians and data collectors).

Blinding:

Trial participants, clinicians, data collectors, and laboratory analysts will be blinded. Blinding of participants and clinicians will be achieved with the use of identical appearing oseltamivir and placebo capsules (achieved via over-encapsulation). Blinding of laboratory technologists is of particular importance since the primary outcome is technologist determined.

Unblinding In the event of a medical emergency, when management of a participant's condition requires knowledge of the study drug, the treatment assignment may be unblinded to disclose the identity of the study drug dispensed. Investigators seeking to unblind the participant's treatment assignment will contact the Principal Investigator (Dr. M. Sholzberg), or in the absence of the Principal Investigator; the Co-Investigator, Dr. Gloria Lim. The Clinical Research Coordinator (CRC) will be contacted to record the reason for unblinding, name of investigator requesting unblinding, date and time of unblinding.

Methods: Data Collection, Management, and Analysis

Source Data The investigators and study staff will maintain adequate and accurate source documentation to document the treatment and study course of a subject and to substantiate the integrity of the trial data submitted for review to regulatory authorities. Documentation will be filled out by study staff and must be completed for each screened subject with all required study data accurately recorded. The investigator has final responsibility for the accuracy and authenticity of the clinical data at all times.

Analysis:

Primary Outcome The primary analysis of platelet glycoprotein will be conducted using ANCOVA where the baseline value is adjusted for. The treatment effect will be expressed as an adjusted mean difference. The intention-to-treat (ITT) approach will be employed for analyses of the primary outcome. If a meaningful difference is observed at day 5 a secondary analysis will employ a linear mixed effect model to explore the duration of the treatment effect.

Secondary Feasibility Outcomes

The investigators have set some minimal targets for the feasibility outcomes that will facilitate assessment of the feasibility to conduct a larger trial. The targets the investigators hope to achieve are:

1. At least 30% of eligible patients recruited
2. Approximately two patients per month recruited
3. At least 80% receive study drug within 12 hours of enrollment
4. At least 90% successful blinding of drug distribution
5. At least 80% completing 12 month follow-up

Secondary Clinical and Biomarker Outcomes Given the small sample size of this trial it must be stressed that all secondary outcomes should be viewed as supportive or describing mechanisms related to the primary findings. Therefore, the statistical methods employed will be used for effect estimation purposes rather than formal statistical inference. The difference in proportion receiving ITP therapy will be expressed as the absolute risk difference with 95% confidence interval. With the exception of the phagocytosis in vitro study (outcome 6), all other biomarkers will undergo a primary analysis of their Day 5 levels. The ANCOVA model will be used to estimated the baseline adjusted difference between groups. If possible (e.g. model convergance) linear mixed effect models will examine the time course of platelets and cytokines by treatment group. In addition to the standard ITT approach, per-protocol analyses of the biomarkers will also be conducted. Finally, "The effects of these antibodies on macrophage- and hepatocyte-mediated Fc-dependent and independent phagocytosis in vitro" is a one-time lab analysis. The difference in mean flourescent intensity will be estimated from a linear regression model that adjusts for antibody class. The possibility of an interaction between treatment and antibody class will also be explored. All biomarker analyses will be supplemented with graphical displays of the results.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age;
* Patients with primary or secondary (i.e. ITP due to a secondary cause) ITP (autoimmune disorder characterized by isolated thrombocytopenia with no other causes or disorders that can be associated with thrombocytopenia; diagnosis of exclusion);
* Individuals with lack of sustained complete remission - platelet count <100 x E9/L despite first line therapy (prednisone, dexamethasone, IVIG);
* Patient's median platelet count over the last 12 months is <100 x E9/L, and must be <100 x E9/L on screening day.

Exclusion Criteria:

* Concurrent medical or surgical treatment for ITP (e.g. prednisone, dexamethasone, IVIG, anti-RhD immune globulin, azathioprine, cyclosporine, cyclophosphamide, danazol, dapsone, mycophenylate mofetil, rituximab, thrombopoietin mimetics, any investigational agents for ITP, splenectomy);
* Patient with a platelet count of <20 x E9/L with active significant bleeding based on a bleeding assessment score of Grade 2 at any site by the ITP Bleeding Scale (IBLS);
* Any immunosuppressive or immunomodulating therapy (not aforementioned) over the last 3 months;
* Oseltamivir therapy over the last 3 months;
* Pregnant females (oseltamivir is a class C drug in pregnancy);
* Lactating females (oseltamivir is detected in low quantities in breast milk).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Mean platelet glycoprotein sialyation | Day 0 and Day 5
  Mean platelet glycoprotein sialyation

SECONDARY OUTCOMES:
Percentage of eligible patients successfully recruited | Screening and Day 0
  Determine the percent of eligible patients that successfully enrolled in the study.
Number of patients recruited per month | Screening and Day 0
  Number of patients recruited per month
Percentage of patients who received the study drug within 12 hours of randomization | Day 0
  Percentage of patients who received the study drug within 12 hours of randomization
Percentage of patients who received every scheduled dose of the study drug in a blinded fashion | Day 0 and Day 5
  Study drug will be dispensed on Day 0 and study drug administration will be assessed on Day 5 by reviewing the blister pack and patient diary
Percentage of patients who had complete follow-up 12 months after randomization | Day 0, Day 5 and Follow up
  Proportion of patients that completed follow-up 12 months after randomization out of the total number of participants that were randomized.
Mean platelet count | Day 0, Day 5 and Follow up
  Mean platelet count
Proportion of patients who received additional ITP based therapy during the study follow-up period | Day 0, Day 5 and Follow up
  Proportion of patients who received additional ITP based therapy during the study follow-up period
Frequencies of CD4+ and CD8+ T regulatory cells | Day 0 and Day 14
  Frequencies of CD4+ and CD8+ T regulatory cells
Cytokine profiles | Day 0 and Day 14
  Cytokine profiles
Anti-platelet glycoprotein antibody specificity/titer | Day 0 and Day 14
  Anti-platelet glycoprotein antibody specificity/titer
Effects of antibodies on macrophage- and hepatocyte-mediated Fc-dependent and independent phagocytosis in vitro | Day 0 and Day 14
  Effects of antibodies on macrophage- and hepatocyte-mediated Fc-dependent and independent phagocytosis in vitro

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, van der Wal DE, Zhu G, Xu M, Yougbare I, Ma L, Vadasz B, Carrim N, Grozovsky R, Ruan M, Zhu L, Zeng Q, Tao L, Zhai ZM, Peng J, Hou M, Leytin V, Freedman J, Hoffmeister KM, Ni H. Desialylation is a mechanism of Fc-independent platelet clearance and a therapeutic target in immune thrombocytopenia. Nat Commun. 2015 Jul 17;6:7737. doi: 10.1038/ncomms8737. PMID 26185093
- [Background] Shao L, Wu Y, Zhou H, Qin P, Ni H, Peng J, Hou M. Successful treatment with oseltamivir phosphate in a patient with chronic immune thrombocytopenia positive for anti-GPIb/IX autoantibody. Platelets. 2015;26(5):495-7. doi: 10.3109/09537104.2014.948838. Epub 2014 Aug 28. PMID 25166956